CLINICAL TRIAL: NCT01471548
Title: A Phase I Dose Escalating Study to Evaluate TKI258 Administered Orally on a 5 Days on/2days Off Schedule in Japanese Patients With Advanced Solid Tumors
Brief Title: Phase I Dose Escalating Study of TKI258
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A1101
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-04

CONDITIONS: Advanced Solid Tumors
Keywords: tumor; cancer; phase1; TKI258
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 (Experimental): dose escalation
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258
  Other Names: Dovitinib

SUMMARY:
The purpose of in this study is to assess the safety profile and estimate the maximum tolerated dose of TKI258 in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures
* Advanced solid tumors
* Agreement to remaining hospitalized
* ECOG performance status of 0 or 1
* Life expectancy of at least 3 months
* Pregnant women. Male and female patients of reproductive potential must agree to employ an effective method of birth control
* Demonstrate the specific hematological /blood chemistry laboratory values

Exclusion Criteria:

* Receipt of any investigational compound within 28 days prior to the first dose of study drug or failure to have recovered from the side effects of such prior therapy
* Receipt of other antineoplastic therapy, including chemo-, hormonal, immuno-, and radiation therapy, within 28 days (with some exceptions)
* Patients with CNS and/or leptomeningeal disease metastases
* Presence or history of thromboembolic or cerebrovascular events
* Impaired cardiac function or clinically significant cardiac disease
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities
* Patients known to be HIV- or HBV- or HCV- positive
* Patients with acute or chronic uncontrolled infection
* Patients who have undergone surgery with general anesthesia for any cause within 28 days prior to the first dose of study drug
* Patients who have been receiving anticoagulant therapy
* Receipt of any hematopoietic colony stimulating factor or blood transfusion within 14 days prior to the first dose of study drug
* Patients who have been administering concomitant medication which may prolong the QTc interval
* Patients with interstitial pneumonia or pulmonary fibrosis proven on a chest CT scan
* Patients with a large volume of ascitic and/or pleural fluid which requires drainage
* Patients with any bone fractures
* Deemed otherwise unsuitable by the investigator

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of TKI258 | 30 days

SECONDARY OUTCOMES:
Antineoplastic activity based on the RECIST criteria | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Hidaka, Saitama

REFERENCES:
- See also: Results for CTKI258A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8745